CLINICAL TRIAL: NCT03814200
Title: A Single-center, Randomized, Double-blind, Two-period Cross-over Study to Investigate the Effect of a Single Intravenous Dose of Rifampicin on the Pharmacokinetics of ACT-246475 in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Rifampicin on the Uptake and Breakdown of ACT-246475 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-076-106; 2018-004226-28 (EudraCT Number)
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Sodium Chloride; selatogrel; Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment period A (Experimental): Treatment A1: saline 0.9%
  followed by
  Treatment A2: ACT-246475
  Interventions: Drug: Saline; Drug: ACT-246475
- Treatment period B (Experimental): Treatment B1: rifampicin
  followed by
  Treatment B2: ACT-246475
  Interventions: Drug: ACT-246475; Drug: Rifampicin

INTERVENTIONS:
Drug: Saline — Single i.v. infusion of 100 mL saline 0.9% for 30 min
  Arms: Treatment period A
Drug: ACT-246475 — Single s.c. dose of 4 mg ACT-246475 in the thigh under fasting conditions
  Other Names: Selatogrel
Drug: Rifampicin — Single i.v. infusion of 600 mg rifampicin (100 mL) for 30 min
  Arms: Treatment period B

SUMMARY:
The study will investigate the effect of rifampicin on the uptake and breakdown of ACT-246475 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure
* Healthy male and female subjects aged between 18 and 65 years (inclusive) at Screening
* Body mass index of 18.0 to 30.0 kg/m2 (inclusive) at Screening
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on the same arm, after 5 min in the supine position at screening and on Day -1 of the first period
* Hematology and coagulation test results not deviating from the normal range to a clinically relevant extent at Screening and on Day -1 of the first period
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day- 1 of the first treatment period and must agree to consistently and correctly use a highly effective method of contraception

Exclusion Criteria:

* Previous exposure to ACT-246475.
* Previous exposure to rifampicin within 3 months prior to Screening.
* Known hypersensitivity to P2Y12 receptor antagonists or rifampicin, or to any of the rifamycins, or any of their excipients
* Loss of 250 mL or more of blood within 3 months prior to Screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol
* Family or personal history of prolonged bleeding (e.g., after surgical intervention) or bleeding disorders (e.g., thrombocytopenia, clotting disturbances), intracranial vascular diseases, stroke, reasonable suspicion of vascular malformations, or peptic ulcers
* Known platelet disorders (e.g., Glanzmann thromboasthenia, von Willebrand disease, platelet release defect)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t) | Up to 36 hours after treatment administration
  The plasma PK parameters of ACT-246475 will be derived by non-compartmental analysis of the plasma concentration-time profiles
AUC from zero to infinity (AUC0-inf) | Up to 36 hours after treatment administration
  The plasma PK parameters of ACT-246475 will be derived by non-compartmental analysis of the plasma concentration-time profiles
The maximum plasma concentration (Cmax) | Up to 36 hours after treatment administration
  The plasma PK parameters of ACT-246475 will be derived by non-compartmental analysis of the plasma concentration-time profiles
The time to reach Cmax (tmax) | Up to 36 hours after treatment administration
  The plasma PK parameters of ACT-246475 will be derived by non-compartmental analysis of the plasma concentration-time profiles
Terminal half-life (t½) | Up to 36 hours after treatment administration
  The plasma PK parameters of ACT-246475 will be derived by non-compartmental analysis of the plasma concentration-time profiles

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schilling U, Dingemanse J, Voors-Pette C, Romeijn C, Dogterom P, Ufer M. Effect of Rifampin-Mediated OATP1B1 and OATP1B3 Transporter Inhibition on the Pharmacokinetics of the P2Y12 Receptor Antagonist Selatogrel. Clin Transl Sci. 2020 Sep;13(5):886-890. doi: 10.1111/cts.12774. Epub 2020 Mar 31. PMID 32166864